CLINICAL TRIAL: NCT04155203
Title: Multi-Center, Double-Blind, Randomized, Vehicle-Controlled, Parallel-Group Study to Compare Perrigo's Mupirocin Cream to A Reference Manufacturer's Mupirocin Cream and to Compare Both Active Treatments to a Vehicle Control in the Treatment of Secondarily Infected Traumatic Skin Lesions
Brief Title: To Compare the Safety and Efficacy of Perrigo's Product to an FDA Approved Product for the Treatment of Secondarily Infected Traumatic Skin Lesions
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Padagis LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: PRG-NY-19-002
Record Dates: First submitted 2019-11-04; First posted 2019-11-07 (Actual); Results first posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Secondarily Infected Traumatic Skin Lesions
MeSH Terms: interventions — Mupirocin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Perrigo active (Experimental)
  Interventions: Drug: Mupirocin Calcium
- Reference Active (Active Comparator)
  Interventions: Drug: Mupirocin Calcium
- Vehicle control (Placebo Comparator)
  Interventions: Drug: Vehicle

INTERVENTIONS:
Drug: Mupirocin Calcium — mupirocin cream
  Arms: Perrigo active
Drug: Mupirocin Calcium — Reference mupirocin cream
  Arms: Reference Active
Drug: Vehicle — vehicle control cream
  Arms: Vehicle control

SUMMARY:
To compare the safety and efficacy of Perrigo's product to an FDA approved product, and to Compare Both Active Treatments to a Vehicle Control in the Treatment of Secondarily Infected Traumatic Skin Lesions

ELIGIBILITY:
Inclusion Criteria:

1. Males or non-pregnant females aged 18 months or older.
2. Must have a secondarily infected traumatic skin lesion such as a laceration, sutured wound, or abrasion.
3. Must have a positive baseline culture for S. aureus and/or S. pyogenes from a sample taken from the secondarily infected traumatic skin lesion.
4. Must have a positive Gram stain or Wright stain for confirmation of white blood cells in the pus/exudate from the secondarily infected traumatic skin lesion.
5. Must have a Skin Infection Rating Scale (SIRS) total score for the secondarily infected traumatic skin lesion of at least 8 at baseline.
6. Must be willing and able to understand and comply with the requirements of the study, apply the medication as instructed, and be able to complete the study.
7. Must be in general good health and free from any clinically significant disease, other than secondarily infected traumatic skin lesion(s), that might interfere with the study evaluations.

Exclusion Criteria:

1. Subjects who are pregnant, breastfeeding, or planning a pregnancy within the period of their study participation.
2. Presence of any dermatological disorder that may interfere with evaluation of the subject's secondarily infected traumatic skin lesion(s).
3. Presence of bacterial skin infection that, because of depth or severity, could not be appropriately treated with a topical antibiotic.
4. Presence of secondarily infected bite or puncture wound.
5. Presence of systemic signs or symptoms of infection (fever defined as an oral temperature greater than 101°F or 38.3°C).
6. Requirement for surgical intervention for treatment of the infection prior to study entry.
7. Presence of cutaneous herpes simplex infections.
8. Use of any topical corticosteroid, topical antibiotic, or topical antifungal, on the secondarily infected target lesion, within 48 hours prior to Visit 1/Day 1.
9. Use of systemic antibiotics or systemic corticosteroids within 7 days of Visit 1/Day 1.
10. Primary or secondary immunodeficiency.
11. Diagnosed Diabetes Mellitus (controlled or uncontrolled).
12. Any uncontrolled, chronic or serious disease or medical condition that would prevent participation in a clinical trial, or, in judgment of the investigator, would put the subject at undue risk or might confound the study assessments.
13. History of hypersensitivity or allergy to mupirocin and/or any ingredient in the study medication.
14. Subject consumes excessive alcohol, abuses drugs, or has a condition that could compromise the subject's ability to comply with study requirements.
15. Subjects who, in the opinion of the investigator, are unlikely to be able to follow the restrictions of the protocol and complete the study.

Min Age: 18 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 657 (Actual)
Dates: Start 2019-10-15 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2021-06-01 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Palm Beach Research Center, West Palm Beach, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Perrigo Active | Reference Active | Vehicle Control
Started | 219 | 219 | 219
Completed | 165 | 184 | 165
Not Completed | 54 | 35 | 54

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Perrigo Active | Reference Active | Vehicle Control | Total
Number analyzed (Participants) | 219 | 219 | 219 | 657
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.58 (16.924) | 20.81 (16.963) | 21.75 (17.089) | 21.38 (16.992)
Age, Customized [Count of Participants; unit: Participants]
  < 18 years old | 100 | 103 | 94 | 297
  18 to 63 years old | 115 | 113 | 120 | 348
  64 to 75 years old | 4 | 3 | 5 | 12
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 96 | 92 | 102 | 290
  Male | 123 | 127 | 117 | 367
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 217 | 219 | 218 | 654
  Not Hispanic or Latino | 2 | 0 | 1 | 3
  Unknown or Not Reported | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 102 | 102 | 102 | 306
  White | 97 | 95 | 93 | 285
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 20 | 22 | 24 | 66

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects in Each Treatment Group With Clinical Cure (Defined as a Skin Infection Rating Scale (SIRS) Score of 0 for All Signs and Symptoms)
Time Frame: 18 days
Measure: Count of Participants; unit: Participants
Arm/Group | Perrigo Active | Reference Active | Vehicle Control
Number analyzed (Participants) | 160 | 181 | 168
Participants | 145 | 169 | 124
Statistical Analysis 1: Comparison: Perrigo Active vs Reference Active; Test type: Equivalence — The primary efficacy endpoint was the proportion of subjects in each treatment group with clinical cure, defined as a SIRS score of 0 for all signs and symptoms at Visit 4/Follow-up (7 days after the end of treatment); equivalence ratio = 0.97, 90% CI 2-sided [-8.19 to 2.70]

ADVERSE EVENTS:
Time Frame: From Day 1 to Day 17
Arm/Group | Perrigo Active | Reference Active | Vehicle Control
All-Cause Mortality (participants affected / at risk) | 0/219 | 0/219 | 0/219
Serious Adverse Events (participants affected / at risk) | 0/219 | 1/219 | 0/219
Other Adverse Events (participants affected / at risk) | 0/219 | 0/219 | 0/219
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Perrigo Active (N=219) | Reference Active (N=219) | Vehicle Control (N=219)
cellulitis (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0) — Cellulitis and abscess of right lower extremity

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2019-02-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT04155203/Prot_000.pdf
  • Statistical Analysis Plan (2021-02-24): https://cdn.clinicaltrials.gov/large-docs/03/NCT04155203/SAP_001.pdf